CLINICAL TRIAL: NCT05115721
Title: A Prospective Study on Establishing the Reference Interval for Pulse Oxygen Saturation in Neonates at High Altitude
Brief Title: Establishing the Reference Interval for Pulse Oxygen Saturation in Neonates at High Altitude
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: Affiliated Hospital of Qinghai University (Other); Qinghai Red Cross Hospital (Other); Qinghai Women and Children's Hospital (Unknown); Geermu People's Hospital (Unknown); Yushu Prefecture People's Hospital (Unknown); Guoluo Tibetan Autonomous Prefecture People's Hospital (Unknown)
Responsible Party: Principal Investigator, Zhangbin Yu, Clinical Professor，Shenzhen People's Hospital, The Second Clinical Medical College of Jinan University
Other Study IDs: NMU-FY2021-59
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: High Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-ductal SpO2
  Interventions: Other: no intervention
- Post-ductal SpO2
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — It's only observational study. No interventions.

SUMMARY:
The now widely used reference interval for pulse oxygen saturation of the neonate after 24 hours of birth has been developed relying on data from low altitude.It is not suitable for neonates at high altitude. At present, no reference interval has been established at high altitude, and the existing studies have many limitations. So this study was designed.

DETAILED DESCRIPTION:
Knowledge of the reference interval of pulse oxygen saturation (SpO2) in neonates is crucial for accurate identification of neonatal hypoxemia. The now widely used standard was derived from low altitude data, which is not suitable neonates at high altitude. At present, many scholars have paid attention to this problem. But, previous studies still have some limitations. For example, they often only focus on a specific altitude. However, with the increase of altitude, the pulse oxygen saturation decreases in a curve, so their study results are only suitable for this specific altitude and can not be widely used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton term infants with no clinical signs and symptoms (e.g., cyanosis, respiratory distress, heart murmur, etc.).

Exclusion Criteria:

* 1. Low birth weight (< 2500 g). 2. Need for oxygen. 3.1 or 5 minute Apgar score < 7. 4. Referred to the neonatal intensive care unit or neonatology department for various reasons. 5. Neonates discharged within 24 hours of birth. 6. Neonates diagnosed with congenital diseases in utero. 7. Refusal of consent.

Ages: 24 Hours to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All consecutively delivered and eligible neonates at the various medical centers at different altitudes during the study will be included. The study period is from November 20, 2021 to November 20, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Pulse oxygen saturation of healthy neonates at high altitude. | 24 hours after birth
  Pulse oxygen saturation of the right hand and any foot of healthy neonates born at high altitude will be measured 24 hours after birth. According to the normality of the results, the distribution range will be described by mean ± standard deviation or range interquartile. Altitude level: ≥ 2000m.

CONTACTS AND LOCATIONS:
Overall Officials: Zhangbin Yu, PHD, Principal Investigator — Jinan University
Locations (1):
- Qinghai Women and Children's Hospital, Xining, Qinghai, China

REFERENCES:
- [Derived] Wang B, Liu C, Yao Y, Lu Z, Yu R, CaiRen Z, Wang Z, Liu R, Wu Y, Yu Z. Establishing the reference interval for pulse oxygen saturation in neonates at high altitudes: protocol for a multicentre, open, cross-sectional study. BMJ Open. 2022 Apr 22;12(4):e060444. doi: 10.1136/bmjopen-2021-060444. PMID 35459680